CLINICAL TRIAL: NCT07326241
Title: Effects of Silver Diamine Fluoride and Intraoral Cryotherapy on Local Anesthesia Efficacy in Permanent Molars With Molar-Incisor Hypomineralization
Brief Title: Effects of Silver Diamine Fluoride and Intraoral Cryotherapy on Local Anesthesia in MIH-Affected Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Burak Carıkcıoglu, Associate Professor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanakkaleOMU4
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: MIH; Molar-Incisor Hypomineralization; Caries Assessment
MeSH Terms: conditions — Molar Hypomineralization | interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Standard Local Anesthesia) (Active Comparator): Standard local anesthesia and operative restorative treatment only (no adjunctive SDF or cryotherapy).
  Interventions: Other: Standard Local Anesthesia
- Intraoral Cryotherapy + Standard Local Anesthesia (Experimental): Intraoral cryotherapy applied before anesthesia, followed by standard local anesthesia and operative restorative treatment.
  Interventions: Other: Standard Local Anesthesia; Other: Intraoral Cryotherapy
- Silver Diamine Fluoride (SDF) + Standard Local Anesthesia (Experimental): Silver diamine fluoride applied before anesthesia, followed by standard local anesthesia and operative restorative treatment.
  Interventions: Other: Standard Local Anesthesia; Other: Silver Diamine Fluoride (SDF)

INTERVENTIONS:
Other: Standard Local Anesthesia — Local anesthesia will be administered using 1.8 mL articaine HCl with 1:100,000 epinephrine (e.g., Ultracain DS) via a standardized block anesthesia technique prior to operative treatment. (Applied in
Other: Intraoral Cryotherapy — Cold application to the buccal mucosa adjacent to the treated tooth for 5 minutes before local anesthetic administration.
  Arms: Intraoral Cryotherapy + Standard Local Anesthesia
Other: Silver Diamine Fluoride (SDF) — SDF will be applied to the target tooth before local anesthetic administration according to standard clinical application procedures.
  Arms: Silver Diamine Fluoride (SDF) + Standard Local Anesthesia

SUMMARY:
Molar-incisor hypomineralization (MIH) is a developmental enamel defect of unclear etiology that affects permanent first molars and often permanent incisors, leading to increased porosity, hypersensitivity, and poor prognosis. The porous structure of MIH-affected enamel facilitates bacterial penetration, which may cause subclinical pulpal inflammation and reduce the effectiveness of local anesthesia during dental procedures. Achieving adequate anesthesia in children with MIH can be challenging, resulting in increased discomfort, anxiety, and behavioral management difficulties.

Cryotherapy has been shown to reduce pain by decreasing local inflammation and slowing nerve conduction, while silver diamine fluoride (SDF) has demonstrated efficacy in reducing dentin hypersensitivity through tubule occlusion, antibacterial activity, and remineralization. This study aims to evaluate the effects of intraoral cryotherapy and silver diamine fluoride application on pain perception and the efficacy of local anesthesia during operative dental procedures in MIH-affected permanent first molars.

DETAILED DESCRIPTION:
The porous enamel structure of MIH-affected teeth facilitates bacterial penetration into enamel and dentin, which may lead to subclinical inflammatory reactions within the dentin-pulp complex. This inflammatory status has been associated with reduced effectiveness of local anesthesia during restorative dental procedures. In pediatric patients, difficulty in achieving adequate anesthesia may result in increased discomfort during treatment, contributing to dental anxiety, negative behavioral responses, and the need for repeated treatment sessions. Therefore, improving anesthetic efficacy in MIH-affected teeth is essential for both patient comfort and treatment quality.

Cryotherapy is a well-established method for pain management in medical practice. Its analgesic effect is attributed to reduced local inflammation, decreased nerve conduction velocity, and minimization of edema and bleeding. Previous studies have demonstrated that the use of cryotherapy following mandibular block anesthesia may reduce pain perception during dental treatment compared to conventional anesthesia alone.

Silver diamine fluoride (SDF) is a solution containing silver and fluoride ions that has been shown to effectively reduce dentin hypersensitivity by occluding dentinal tubules, promoting remineralization of demineralized tooth structure, and exerting antibacterial effects. SDF stabilizes active carious lesions and reduces sensitivity through the formation of fluorohydroxyapatite and tubule blockage. It was approved by the U.S. Food and Drug Administration in 2014 for the treatment of dentin hypersensitivity. Given its desensitizing properties, SDF may be a promising adjunctive approach to enhance anesthetic effectiveness in MIH-affected molars.

This study aims to evaluate the effects of intraoral cryotherapy and silver diamine fluoride application on pain perception and the efficacy of local anesthesia during operative dental procedures in permanent first molars affected by MIH. Pediatric patients presenting for examination and treatment at the Department of Pediatric Dentistry will be allocated into three groups: a control group, a cryotherapy group, and an SDF group. Prior to treatment, demographic and dental characteristics will be recorded, and baseline pulp sensibility responses will be assessed using electric cold testing and air stimulation (SCASS).

All treated teeth will receive local anesthesia using a standardized mandibular block technique. In the SDF group, SDF will be applied prior to anesthetic administration. In the cryotherapy group, cold application will be performed on the buccal mucosa for 5 minutes using frozen saline contained in 2-mL dental syringes wrapped in sterile gauze before treatment. Following local anesthesia, caries removal and final composite resin restorations will be completed. Pain intensity and behavioral responses during treatment will be assessed using validated pediatric pain scales. The total duration of the clinical procedure is planned to be approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 12 years.
* Systemically healthy children with no medical conditions that could interfere with dental treatment.
* Presence of at least one permanent first molar affected by molar-incisor hypomineralization (MIH), diagnosed according to the European Academy of Paediatric Dentistry (EAPD) criteria.
* Teeth with caries lesions classified as ICDAS II codes 2, 3, 4, 5, or 6.
* Children with an adequate level of cooperation to allow completion of dental treatment under clinical conditions.
* Children and their parents/legal guardians who have read, understood, and signed the informed consent form and agreed to participate in the study.

Exclusion Criteria:

* Teeth that are not restorable.
* Children with a known allergy or hypersensitivity to any materials used in the study, including local anesthetics, silver diamine fluoride, or restorative materials.
* Presence of spontaneous pain, percussion sensitivity, or other signs/symptoms of pulpal pathology in the study tooth.
* Children with systemic diseases or conditions that could affect pain perception, healing, or cooperation during dental treatment.
* Children who are unable or unwilling to complete the clinical procedure.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during dental treatment (FLACC) | Immediately after completion of the dental procedures
  Face, Legs, Activity, Cry, Consolability scale will be recorded. Each category is scored on the 0 to 2 scale. Add the scores together (for a total possible score of 0 to 10).
Pain intensity during operative dental treatment (Wong-Baker) | Immediately after the dental procedures were completed
  The patient's current pain was assessed using the Wong-Baker Faces Pain Rating Scale, with scores ranging from 0 to 5, where higher scores indicate greater pain intensity and a worse outcome, and the assessment was performed immediately after completion of the dental procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Çarıkçıoğlu, Associate Professor, Principal Investigator — Çanakkale Onsekiz Mart University; Seçkin Aksu, Assistant Professor, Study Director — Mersin University; Hilal Öztürk, Research Assistant, Study Chair — Çanakkale Onsekiz Mart University
Locations (2):
- Turkey (Türkiye) (2):
  - Çanakkale Onsekiz Mart University, School of Dentistry, Çanakkale
  - Mersin University, School of Dentistry, Mersin

IPD SHARING:
Plan to Share IPD: Undecided